CLINICAL TRIAL: NCT04932915
Title: A Randomized Placebo-controlled Phase 2 Study to Assess the Safety and Efficacy of UNI91103 Intranasal Administration in Adults With Asymptomatic or Mildly Symptomatic COVID-19
Brief Title: Safety and Efficacy of Intranasal Administration of Niclosamide (UNI91103) in Adults With Asymptomatic or Mild COVID-19
Acronym: PREVENT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Failure of recruiting patients
Sponsor: UNION therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNI91103-201; 2021-001036-25 (EudraCT Number)
Record Dates: First submitted 2021-06-18; First posted 2021-06-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Niclosamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UNI91103 intranasal spray 1% (Experimental): UNI91103 intranasal spray 1%, BID, 10 consecutive days
  Interventions: Drug: Niclosamide
- Placebo (Placebo Comparator): Placebo intranasal spray, BID, 10 consecutive days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide — Niclosamide is a broad spectrum, host targeting antiviral that inhibits viral replication (by neutralizing endosomal pH) and increases viral clearance (by increasing the autophagic flux). The niclosamide solution is administered directly to the nasal cavity via a nasal spray.
  Arms: UNI91103 intranasal spray 1%
Drug: Placebo — The placebo formulation contains purified water, sodium chloride as common isotonizing agent and the FAO/WHO approved colorant FD&C Red 40 to match the red-orange colour of the active solution. The solution is administered directly to the nasal cavity via a nasal spray.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of UNI91103 intranasal spray for treatment of coronavirus disease 2019 (COVID-19) in asymptomatic or mildly symptomatic adults.

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female aged ≥45 and <80 years
* Subject is tested to confirm infection with SARS-CoV-2 on a sample taken within 3 days before randomization
* Subject is either without symptoms or has 1 or more of the following symptoms: Stuffy or runny nose, Sore throat, Loss of taste, Loss of smell, Headache.

None of the symptoms should have been present >5 days.

Exclusion Criteria:

* Subject has an underlying condition that may interfere with intranasal administration of the IMP (e.g., chronic ulcers in the nose).
* Subject has symptoms suggesting engagement of the lower respiratory tract or a systemic engagement
* Subject has an active or acute infection other than SARS-CoV-2
* Subject has another member of the same household recruited to this study

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-09-03 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with worsened symptoms any time from Day 3 to Day 10 compared with baseline | Day 3 to Day 10
  Worsening is assessed by the Food and Drug Administration (FDA) COVID-19 Symptom Questionnaire, assessing severity of symptoms over the past 24 hour period.

SECONDARY OUTCOMES:
Proportion of subjects with worst intensity/grade up to Day 10 and up to Day 15 in any single symptoms in the 3 domains of the FDA COVID-19 questionnaire | Day 10 and up to Day 15
  Assessed by the FDA COVID-19 symptom questionnaire divided into 3 domains - Items 1 to 10, items 11 to 12 and items 13 to 14
Proportion of subjects reporting the following number of symptoms with worst intensity/severe grade: ≥ 1 symptom, ≥ 2 symptoms, ≥ 3 symptoms, etc. | Any time point
  Assessed by the FDA COVID-19 symptom questionnaire looking at the individual symptoms
Proportion of subjects with worsened symptoms at Day 15 compared with baseline. | Day 15
  Worsening is assessed by the FDA COVID-19 Symptom Questionnaire, which is a self reported questionnaire assessing severity of symptoms over the past 24 hour period.
Change from baseline in each single symptom score | Days 10, 15 and 30
  Assessed by the FDA COVID-19 symptom questionnaire looking at the individual symptoms
Proportion of subjects who are asymptomatic on Day 10 | Day 10
  Assessed by the FDA COVID-19 symptom questionnaire
Proportion of subjects requiring visits to urgent care (UC) or emergency department (ED) facilities, or hospitalization because of signs or symptoms of COVID-19 | Day 10, 15 and 30
  Number of visits to urgent care (UC) or emergency department (ED) facilities, or hospitalization is assessed by a self developed questionnaire
Proportion of subjects admitted to intensive care units (ICU) and/or died | At screening, Day 1, and every other day through Day 10, and again at Day 15 and Day 30
  Assessed by WHO 11-point Ordinal Scale
Change from baseline in SARS-CoV-2 viral load at Day 5 and Day 10 | Day 5 and Day 10
  Assessed by quantitative reverse transcription polymerase chain reaction (qRT-PCR)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Heymer, MD, Principal Investigator — Klinische Forschung Dresden GmbH
Locations (3):
- Germany (3):
  - Klinische Forschung Berlin-Mitte GmbH, Berlin
  - Klinische Forschung Dresden GmbH, Dresden
  - Klinische Forschung Hamburg GmbH, Hamburg

IPD SHARING:
Plan to Share IPD: No